CLINICAL TRIAL: NCT05463549
Title: The Effect of Exposure to an Informative Video About Amniocentesis Before the Procedure on Maternal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0169-21-WOMC
Record Dates: First submitted 2022-03-27; First posted 2022-07-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Related; Anxiety in Pregnancy; Amniocentesis Affecting Fetus or Newborn
Keywords: explanatory video; anxiety reduction; amniocentesis; pregnancy

STUDY DESIGN:
Intervention Model Description: Women assigned to undergo amniocentesis during the trail time-period will be invited to participate in the study and will be signed a consent form.The randomization will be based on different days for each intervention - a day specified to women comprising of the research group while the following clinic day will be dedicated to women from the control group.
  The study group will watch an informative video while waiting for amniocentesis, and the control group will not watch the video while waiting.
Who Masked: Outcomes Assessor
Masking Description: Data regarding maternal characteristics, anxiety and pain levels as reported by the patients via the questioners will be stored according to random serial numbers without intervention type. The investigator handling the statistical analysis will be unaware of the patient's exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informative video (Experimental): The research group will be exposed to an informative instructional film before the procedure.
  Interventions: Other: Informative video
- No video (No Intervention): The control group will undergo amniocentesis with information given as accepted by standard-of-care.

INTERVENTIONS:
Other: Informative video — An informative instructional film regarding the amniocentesis procedure including answers to frequently asked questions.
  Arms: Informative video

SUMMARY:
The effect of exposure to an informative video about amniocentesis before the procedure on maternal anxiety

DETAILED DESCRIPTION:
Amniocentesis is a common sonography-guided procedure that is usually preformed during the second trimester of pregnancy in order to obtain neonatal genetic information. Previous studies have shown that although the risk of a major complication is small, many women experience profound anxiety regarding the procedure.

Many stress-relieving techniques have been proposed and studied concerning stress-related interventions during pregnancy. However, the use of an informative video that is a simple, accessible, widely accepted tool has not been tested in the context of amniocentesis. In this interventional study the investigators aim to examine the effect of an informative pre-procedural video on anxiety and pain levels in women undergoing amniocentesis.

ELIGIBILITY:
Inclusion Criteria:

* Women who come for amniocentesis in the Edith Wolfson Medical Center
* Women who sign a consent form to enroll to the study.

Exclusion Criteria:

* Women under 18 years of age.
* Women who do not speak Hebrew

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of change in anxiety levels between before and after undergoing the amniocentesis | Each patient will answer the STAI questionnaire twice - within 2 hours before the operation and watching the video (S1) and within 30 minutes after performing amniocentesis (S2) to assess the change in anxiety levels before and after the operation
  Women recruited to the study will answer the Spielberger's state-trait anxiety inventory questionnaire- a validated questionnaire for assessing anxiety which includes 20 statements expressing different states of anxiety. The patients will be asked to rate to what extent they currently relate to the statement written on a scale of 1 to 4 (1- does not agree at all and 4- strongly agrees). The final score in each questionnaire is obtained by summing the scores of each statement, while the scores of positive statements reflecting anxiety-free behavior will be reversely summed. Higher scores indicate higher level of anxiety.

SECONDARY OUTCOMES:
Intensity of pain, discomfort, satisfaction with the video and satisfaction in general | The questionnaire will be filled within 30 minutes after performing amniocentesis
  These parameters will be measured using the item visual analog scales 11 questionnaire containing questions reflecting pain, discomfort and satisfaction levels. Each statement scores between 0-10 as a reflection of the patients' identification with the statement- each statement reflecting different aspects of the patients' experience:
  question 1- pain during the procedure question 2- pain 10 minutes after the procedure question 3- general unpleasantness question 4- anxiety during procedure question 5- satisfaction with information about procedure question 6- overall satisfaction with treatment question 7- level of discomfort as a result of informative video prior to the amniocentesis question 8- level of anxiety caused by watching the informative video question 9-importance of informative video for understanding the amniocentesis procedure

CONTACTS AND LOCATIONS:
Overall Officials: Or Marom, Dr, Principal Investigator — Edith Wolfson Medical center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: Yes
Unidentified patient data will be shared between researchers for statistical analysis, other unidentified data will be published.
Supporting Information: Study Protocol, SAP
Time Frame: Within the first 5 years from publication.
Access Criteria: Researches in need of data will request permission from study organizers by mail including data needed, purpose of data sharing and data protection steps.

REFERENCES:
- [Derived] Marom O, Weiner E, Gindes L, Mor L, Gury M, Toledano E, Alon AS, Miremberg H, Shalev J, Levy M. The effect of watching an informational video prior amniocentesis on maternal anxiety: a randomized controlled trail. Arch Gynecol Obstet. 2024 Aug;310(2):1001-1008. doi: 10.1007/s00404-023-07288-y. Epub 2023 Dec 7. PMID 38060016